CLINICAL TRIAL: NCT02446093
Title: Neoadjuvant CAN-2409 Plus Prodrug in Combination With Chemoradiation or Stereotactic Body Radiation Therapy for Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: Neoadjuvant CAN-2409 in Combination With Chemoradiation or SBRT for Borderline Resectable Pancreatic Adenocarcinoma
Acronym: PaTK02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PaTK02
Record Dates: First submitted 2015-04-14; First posted 2015-05-18 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2023-05

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma
Keywords: Borderline resectable pancreatic adenocarcinoma; Immunotherapy; Aglatimagene besadenovec; Neoadjuvant; CAN-2409
MeSH Terms: interventions — Chemoradiotherapy; Radiosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Arm (Experimental): CAN-2409 + prodrug (valacylovir or acyclovir) in combination with neoadjuvant chemoradiation or SBRT + Surgery
  Interventions: Biological: Aglatimagene besadenovec; Radiation: Chemoradiation; Radiation: Stereotactic body radiation therapy; Procedure: Surgery
- Control Arm (Active Comparator): Neoadjuvant chemoradiation or SBRT + Surgery
  Interventions: Radiation: Chemoradiation; Radiation: Stereotactic body radiation therapy; Procedure: Surgery

INTERVENTIONS:
Biological: Aglatimagene besadenovec — Three courses of CAN-2409 + prodrug (valacylovir or acyclovir) will be delivered and timed with different phases of therapy: 1) after induction chemotherapy 2) during CR or post-SBRT, and 3) at time of surgery. Up to 2 additional courses of CAN-2409 + prodrug, if feasible, for subjects with disease progression or metastases.
  Other Names: CAN-2409; AdV-tk
  Arms: Test Arm
Radiation: Chemoradiation — CR will start not more than 2 months after completion of induction chemotherapy. The chemotherapy component of CR may be selected as per institutional standard of care (SOC) and protocols for administration, and may include capecitabine, 5-FU, or gemcitabine. Radiation should consist of a total dose of 45-54 Gy in 1.8-2.0 Gy fractions concurrent with chemotherapy over 3-5.5 weeks.
Radiation: Stereotactic body radiation therapy — SBRT should start no more than 2 months after completion of induction chemotherapy. For SBRT, the radiation should consist of a total dose of 25-50 Gy in divided fractions over 1-2 weeks.
Procedure: Surgery — Surgical resection should be performed within 8 weeks after completing CR or SBRT.

SUMMARY:
The purpose of this study is to characterize the safety, preliminary efficacy, and immune biologic activity of CAN-2409 + prodrug (valacyclovir or acyclovir) in subjects with borderline resectable pancreatic cancer who are being treated with neoadjuvant chemoradiation (CR) or stereotactic body radiation therapy (SBRT). The Standard of Care (SOC) Control arm will be used as a benchmark for informal comparisons of efficacy, safety, and biomarkers.

DETAILED DESCRIPTION:
Study design is an open-label Phase 2 trial that randomizes subjects with borderline resectable pancreatic adenocarcinoma to received SOC with (Test arm) or without (Control arm) the addition of CAN-2409 + prodrug (2:1 randomization, Test: Control), beginning after completion of at least 4 months (8 cycles) of a FOLFIRINOX based induction therapy. Confirmation of borderline resectable status will be based on central radiologic review following completion of FOLFIRINOX based induction regimen. Upon enrollment, eligible subjects will receive three courses of CAN-2409 + prodrug, the first course starting prior to CR or SBRT, the second course concurrent with CR or just following completion of SBRT, and the third at time of resection. Up to 2 additional courses are allowed at the time of disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of pancreatic adenocarcinoma adequately treated with a FOLFIRINOX based induction chemotherapy for at least 4 months such that they are a candidate for localized therapy with CR or SBRT followed by surgery with or without major vascular resection.
2. Subjects must be deemed to be in adequate health to undergo major surgery (e.g., pancreaticoduodenectomy).
3. Tumor accessible for injection by EUS or CT-guidance, considered potentially resectable at time of diagnosis, and classified as borderline resectable based on central radiologic review of CT scans performed following completion of FOLFIRINOX based induction chemotherapy. Resection may include major vascular resection with reconstruction as needed.

   Criteria for borderline resectable disease status:
   * No distant metastasis or lymph node involvement outside the planned resection field.
   * Venous involvement of the superior mesenteric vein (SMV) or portal view (PV) with distortion or narrowing of the vein or occlusion of the vein with suitable vessel proximal and distal, allowing for safe resection and replacement
   * Gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct tumor abutment of the hepatic artery, without extension to the celiac axis
   * Tumor abutment of the superior mesenteric artery (SMA) not to exceed > 180 degrees of the circumference of the vessel wall
4. Age > 18 years at the time of consent
5. Performance status ECOG 0 or 1
6. SGOT (AST) <3x upper limit normal
7. Total bilirubin <2mg/dl

   * Subjects with biliary obstruction can be enrolled if AST and bilirubin do not meet criteria but must meet the criteria after stenting before starting treatment
8. Creatinine <2mg/dl
9. Calculated creatinine clearance > 30ml/min
10. WBC > 3000/mm^3
11. Absolute neutrophil count (ANC) > 1000/mm^3
12. Platelets > 100,000/mm^3
13. Hemoglobin > 9g/dl
14. Signed, written informed consent

Exclusion Criteria:

1. Primary hepatic dysfunction including known cirrhosis or active hepatitis. Subjects with biliary obstruction must be stented prior to initiating treatment
2. Evidence of clinically significant pancreatitis as determined by the investigator
3. Evidence of significant ascites as determined by investigator
4. Subjects on systemic corticosteroid (>10 mg prednisone per day or equivalent), systemic immunomodulators, or other systemic immunosuppressive drugs
5. Known to be HIV+
6. Pregnant or breast-feeding. Female subjects of childbearing age must have negative serum or urine pregnancy test within 2 weeks of beginning protocol therapy
7. Other current malignancy (except squamous or basal cell skill cancers)
8. Other serious co-morbid illnesses or compromised organ function
9. Known sensitivity or allergic reactions to acyclovir or valacyclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-10; Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety grade by CTCAE version 4.0 | From the time of CAN-2409 administration to 30 days after the last dose of valacyclovir.
  Frequency of adverse events.
Survival Rate | 24 months
  All eligible subjects will be followed for at least 2 additional years from the completion of primary treatment window.

SECONDARY OUTCOMES:
Overall survival (OS) from time of diagnosis | 60 months
  Time from diagnosis until death from any cause.
Overall survival (OS) from time of study enrollment | 60 months
  Time from enrollment until death from any cause.
Progression free survival (PFS) from time of diagnosis | 60 months
  Time from diagnosis until first objective documentation of progression (local or distant) or death from any cause.
Progression free survival (PFS) from time of study enrollment | 60 months
  Time from study enrollment to documented disease progression or death from any cause.
Resection rate | 12 weeks
  Subjects will be considered to have R0 resection if all lesions are removed with negative microscopic surgical margins. Subjects will be considered to have R1 resection if all lesions are removed with any positive microscopic surgical margins.
Disease free survival (DFS) in subjects with R0 resection | 60 months
  Disease-free survival (DFS) will be measured from R0 resection until first objective documentation of recurrence or death from any cause.
Immunological biomarker characterization in tumor and peripheral blood | 24 months
  Immunophenotyping in the blood and in the tissue.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Lee Health/Regional Cancer Center, Fort Myers, Florida
  - Ohio State University, Columbus, Ohio
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico